CLINICAL TRIAL: NCT06938022
Title: Chronic Airway Inflammation: The Impact of Respiratory Microbiota, Infection Characteristics, and Imaging Features on Disease Progression and Quality of Life-A Multomic and Comprehensive Study
Brief Title: Respiratory Microbiota, Infection Characteristics and Imaging Manifestations in Patients With Chronic Airway Inflammation
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Other Study IDs: 2025-108A-01
Record Dates: First submitted 2025-03-31; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Chronic Airway Inflammation; Asthma; Chronic Obstructive Pulmonary Disease; Bronchiectasis
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- ICS treatment sensitivity and resistance in Chronic Airway Inflammation: Using a prospective, single-center, observational study design, 240 patients were planned to be enrolled, divided into ICS-sensitive and resistant. Through multi-omics technologies such as 16S rRNA gene sequencing, metagenomic sequencing, and metabolomics analysis, the composition, structure and functional gene differences of airway and intestinal microbiota were analyzed, and the microbiota-metabolite-host network was constructed by combining inflammatory factor detection and transcriptomic analysis, and the complex mechanism of ICS treatment response was analyzed.
- The study of respiratory viral infection and inflammatory markers in patients with acute exacerbatio: A prospective, open-label, self-controlled trial design was adopted, and 150 patients were expected to be included. RT-PCR was used to detect respiratory viruses, and ELISA was used to detect inflammatory markers, and the dynamic changes of viral infection and inflammatory markers and their association with clinical phenotypes were analyzed.
- The effect of respiratory viral infection on the airway inflammation and disease severity of asthma: Patients aged 18-80 years with a clinical diagnosis of asthma exacerbation were included, nasopharyngeal swabs and sputum samples were collected for viral analysis, and ELISA was used to detect airway inflammation markers, and the number and severity of acute exacerbations, hospitalization and questionnaire scores were evaluated.
- The clinical significance of fungal infection in acute exacerbation of bronchiectasis: A prospective, observational study design was used and 150 patients were expected to be included. The diversity and abundance of fungi in sputum were detected by 18S rRNA technology, and the inflammatory markers were detected by ELISA, and the relationship between fungal infection and clinical manifestations, questionnaire scores and inflammatory markers was analyzed.
- The role of pulmonary function test and chest CT in predicting acute exacerbation of chronic obstruc: A prospective, observational cohort study design was adopted, and 200 patients were expected to be included. Pulmonary function tests, bronchodilator tests, chest CT scans, etc., were followed up for 1 year, and the changes in symptoms, acute exacerbations and all-cause mortality were recorded, and the biomarkers predicting acute exacerbations were analyzed using statistical models.
- The predictive value of baseline pulmonary function and radiomics in acute exacerbation of bronchiec: A prospective, observational clinical trial design is adopted, and 150 patients are expected to be included. The clinical data, pulmonary function indexes and thin-slice CT scan results of the patients were collected, and the follow-up was 1 year, and the number of acute exacerbations, hospitalization and quality of life scores were recorded for statistical analysis.

SUMMARY:
This study，Respiratory microbiota, infection characteristics and imaging manifestations in patients with chronic airway inflammation， adopted a prospective, observational, multi-omics study design to comprehensively evaluate the effects of respiratory microbiota, infection characteristics and imaging manifestations on disease outcomes and quality of life in patients with chronic airway inflammation. Involving six parallel sub-studies, These include: (1) the differences and mechanisms of lung microecology in ICS treatment sensitivity and resistance in patients with chronic airway inflammation, (2) the study of respiratory viral infection and inflammatory markers in patients with acute exacerbation of chronic obstructive pulmonary disease, (3) the effect of respiratory viral infection on the airway inflammation and disease severity of asthma in acute exacerbation, (4) the clinical significance of fungal infection in acute exacerbation of bronchiectasis, (5) the role of pulmonary function test and chest CT in predicting acute exacerbation of chronic obstructive pulmonary disease, and (6) the predictive value of baseline pulmonary function and radiomics in acute exacerbation of bronchiectasis， Each sub-study targeted a different study purpose and a specific patient population. All sub-studies followed uniform research principles, including scientificity, ethics, and consistency. All subjects were required to sign an informed consent form before enrollment to ensure that they understood the purpose, process, possible risks and privacy protection measures of the study. The study plans to enroll about 1,000 eligible patients covering chronic airway inflammatory diseases such as asthma, chronic obstructive pulmonary disease (COPD) and bronchiectasis.

In this study, multi-omics techniques, including microbiome, metabolomics, radiomics, and transcriptomics, were used to comprehensively evaluate the effects of respiratory microbiota, infection characteristics, and imaging manifestations on disease outcomes and quality of life in patients with chronic airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

(1) Age: 18 to 80 years old (inclusive), without restrictions on gender or ethnicity.

(2) Disease Diagnosis:

1. COPD patients must meet the GOLD diagnostic criteria, with post-bronchodilator FEV1/FVC < 70% and FEV1 < 80% of the predicted value.
2. Asthma patients must meet clinical diagnostic criteria, including recurrent wheezing, shortness of breath symptoms, frequently occurring at night; during attacks, wheezing sounds can be heard in both lungs; effective treatment with bronchodilators or corticosteroids, or symptoms can be relieved spontaneously, and at least one of the following tests must be positive: positive bronchial provocation test; positive bronchodilator test with FEV1 increase ≥12%, and FEV1 increase absolute value ≥200ml; daily peak expiratory flow (PEF) variability ≥10% within one week.
3. Bronchiectasis patients must meet the diagnostic criteria based on CT imaging, including: bronchial diameter/accompanying pulmonary artery diameter ratio >1; high-resolution CT (HRCT) showing dilated cystic, columnar, or cystic bronchial shadows.

(3) Disease Status:

1. Patients with chronic airway inflammation must be in a stable phase, defined as no acute exacerbations, hospitalizations, or use of other treatments for at least 4 weeks.
2. COPD patients with acute exacerbations must meet the definition of acute exacerbation: at least two major symptoms (dyspnea, increased sputum, and purulent sputum) worsen, or at least one major symptom and one minor symptom (wheezing, sore throat, cough without other causes, and fever) worsen.
3. Asthma patients in the acute attack phase must meet the definition of acute attack: sudden worsening of symptoms (including wheezing, shortness of breath, chest tightness, cough, etc.), decreased lung function, poor response to routine treatment, other clinically diagnosed acute attacks.
4. Bronchiectasis patients with acute exacerbations must meet the definition of acute exacerbation: increased cough, increased sputum or sputum viscosity, purulent sputum, dyspnea or decreased exercise tolerance, fatigue or discomfort, hemoptysis, at least three of the above six symptoms occur newly or significantly worsen, lasting ≥48 hours.

(4) Treatment Status:

1. In the chronic airway inflammation patient ICS treatment study, patients must require ICS treatment under routine care, i.e., have been recommended to use ICS and are currently using ICS treatment.
2. In other studies, patients must maintain unchanged long-term medication during the follow-up period, but may be appropriately adjusted according to the attending physician's clinical decision.

(5) Others:

1. All participants must voluntarily participate in the study and sign the informed consent form.
2. Patients must be able to communicate in language or writing, understand and sign the content of the informed consent form, and be able to complete the required pulmonary function and other auxiliary examinations for the trial.

Exclusion Criteria:

(1) Recent Medication Use:

1. In the chronic airway inflammation patient ICS study, exclude patients who have used corticosteroid-related treatment within the last 3 months, exclude patients who have received antibiotic treatment within the last 3 months.
2. In other studies, exclude patients who have used antibiotics, immunosuppressants, cytotoxic agents, or hormones systemically within the last 4 weeks.

(2) Other Significant Diseases:

1. Clinically significant pulmonary diseases other than the study disease, such as active tuberculosis, pulmonary embolism, pneumothorax, pneumothorax, pulmonary hypertension, interstitial lung disease, lung cancer, pulmonary fibrosis, tuberculosis, etc.
2. Severe other systemic diseases, such as myocardial infarction, severe arrhythmia, liver dysfunction, renal insufficiency, rheumatic immune system diseases, hematological diseases, active malignant tumors, etc.

(3) Disease Status:

[1] Patients who have experienced any degree of acute exacerbation within the last 4 weeks before screening for the stable phase study.

(4) Special Populations:

1. Female patients who are pregnant or breastfeeding.
2. Patients with poor compliance.
3. Patients who cannot complete sample collection due to physical or psychological factors, especially those who need to collect multiple samples.
4. Patients who are participating in other clinical trials. (5) Related Contraindications:

[1] Patients with contraindications to pulmonary function tests and chest CT, such as chest metal, history of myocardial infarction, stroke, aortic aneurysm, or ocular surgery or retinal detachment within the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical diagnosis of chronic airway inflammation (including COPD, asthma, and bronchiectasis), aged 18-80 years, meeting the inclusion criteria and having no exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory microorganisms | Baseline, Week 4 (mid-intervention), and Week 8 (end of intervention) follow-up.
  Multiplex RT-qPCR analysis was performed to analyze the microbial species and abundance of respiratory tract microorganisms in sputum samples, nasopharyngeal swabs or exhaled air condensate of patients with chronic airway inflammation
ACT（Asthma Control Test） Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  In the research group of ICS treatment sensitivity and resistance in Chronic Airway Inflammation, Asthma symptom control will be assessed using the Asthma Control Test (ACT), a validated questionnaire with scores ranging from 5 to 25. Higher scores indicate better asthma control.
CAT（COPD Assessment Test） Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  In the research group of ICS treatment sensitivity and resistance in Chronic Airway Inflammation, Chronic Obstructive Pulmonary Disease Assessment Test（CAT) is a tool used to assess the severity of chronic obstructive pulmonary disease (COPD) and the quality of life of patients. The scoring range is 0 - 10 points. Grade division: 0 - 2 points: Mild. 3 - 5 points: Moderate. 6 - 10 points: Severe.

SECONDARY OUTCOMES:
Changes in Airway Inflammation Markers | Baseline, Week 4, Week 8 follow-up.
  Detection of airway inflammatory factors by ELISA, such as IL-4, IL-5, IL-6, IL-8, IL-13, IL-33, TNF-α, IL-1β, etc.The concentration of Airway Inflammation Markers is measured in pg/mL.
FEV1（Forced Expiratory Volume in 1 second） | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  Pulmonary function FEV1 index was evaluated in liters (L). It refers to the volume of air exhaled in the first second by the subject exhaling at the fastest rate after the maximum inspiration.
PEF（Peak Expiratory Flow） | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  PEF is measured in liters per minute (L/min). It refers to the maximum flow rate that can be achieved when exhaling at the fastest speed after the maximum inspiration. This indicator can reflect how open the airway is.
MMEF75/25（Maximal Mid-Expiratory Flow between 75% and 25% of FVC） | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  MMEF75/25 is measured in liters per minute (L/min). This is the average expiratory flow rate over the course of 75% to 25% of the forced expiratory volume. It is primarily used to assess the function of the small airways.
FVC（Forced Vital Capacity） | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  FVC is measured in liters (L). It is the maximum volume of air that can be exhaled by exhaling forcefully as fast as possible after the maximum inhalation. This indicator reflects the ventilatory function of the lungs. FVC is generally around 3.5 - 5 L in normal adult males and slightly lower in females. FVC can be used to assess the elasticity of the lungs, the patency of the airways, etc.
FEV1/FVC（Forced Expiratory Volume in 1 second to Forced Vital Capacity Ratio） | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  The unit of FEV1/FVC is %. It is mainly used to determine if there is an airflow obstruction. Normally, FEV1/FVC should be greater than 70%.
Blood Routine Test | Baseline, Week 4 , Week 8 follow-up.
  Including CRP, WBC, Neu, Mono, Eos, RBC, Hb, and PLT.
Serum viral Antibody IgG | Baseline, Week 4 , Week 8 follow-up.
  The serum viral antibody titer is measured by ELISA, which is a commonly used method for detecting and quantifying antibodies in patient samples. Then, these results will be used to analyze the relationship between viral infection and disease status, severity, or treatment response.
Anxiety Levels | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  Anxiety symptoms will be assessed using the Hamilton Anxiety Rating Scale (HAMA), a validated scale with scores ranging from 0 to 56, where higher scores indicate greater anxiety severity.
Depression Levels | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  Depressive symptoms will be observed using the Hamilton Depression Rating Scale (HAMD), which scores from 0 to 52, with higher scores indicating more severe depression.
Incidence of Serious Adverse Events (SAEs) | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  The safety will be assessed by monitoring and recording the incidence of treatment-emergent serious adverse events (SAEs) using the Serious Adverse Event Report Form (SAE Report). The research team will document, analyze, and provide appropriate medical responses to any incidents.
Number of Emergency Visits and Hospitalizations | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  Record the number of emergency visits and hospitalizations to evaluate the clinical effectiveness of treatment.
Number of Acute Exacerbations | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  The unit of Number of Acute Exacerbations is number of events. Total count of acute exacerbations experienced by participants.
Exacerbation Events | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  Acute exacerbation events of the disease will be assessed using Asthma, COPD, Bronchiectasis exacerbation records, recording the timing, frequency, and severity of each exacerbation. and grade the severity as mild, moderate, or severe.
Frequency of Emergency Department Visits | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  The number of emergency department visits due to acute exacerbations of Asthma, Chronic Obstructive Pulmonary Disease (COPD), and Bronchiectasis will be tracked using patients' self-reports and verified through medical records. This measure helps to evaluate the severity of the diseases.
Frequency of Hospitalizations | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  The number of people hospitalized due to acute exacerbations of Asthma, COPD (Chronic Obstructive Pulmonary Disease), and Bronchiectasis will be recorded, including detailed information such as the length of hospital stay and the treatments administered.
Severity Grading of Acute Exacerbations | Baseline, Week 4, Week 8, 3-month, 6-month, 9-month, and 12-month follow-up.
  The unit of Severity Grading of Acute Exacerbations is units on a severity scale. Severity of each acute exacerbation categorized by a standardized scale (e.g., mild/moderate/severe or graded numerically, such as Grade 1-3).
Occurrence of Respiratory Failure | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  Documentation of respiratory failure events during hospital stays, including clinical criteria for diagnosis and management details.
Number of Moderate to Severe Acute Exacerbations | Baseline, Week 4, Week 8, 3-month, 6-month, 9-month, and 12-month follow-up.
  The unit of Number of Moderate to Severe Acute Exacerbations is number of events. Count of exacerbations classified as moderate or severe based on the severity grading scale.
Use of Non-Invasive Ventilation | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  Documentation of the use of non-invasive ventilation during hospitalization, including indications and duration of use.
ICU Admission and Intubation | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  Records of ICU admissions and whether intubation was required during hospitalization, including associated clinical details.
Systemic Steroid Use | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  Documentation of systemic corticosteroid use during hospital stays, including dosage and duration.
Length of Hospital Stay | Baseline, Week 4, Week 8，3-month，6-month，9-month，and 12-month follow-up.
  Total duration of each hospital stay will be recorded to assess the impact of the intervention on hospitalization length.
CAT（COPD Assessment Test） Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  It is used to evaluate the quality of life of COPD patients in groups other than the chronic airway inflammation ICS research group. It includes 8 items, involving dyspnea, exercise ability, cough, sputum, chest tightness, sleep quality, self - confidence and energy level. The scoring range is 0 - 10 points.
  Grade division:
  0 - 2 points: Mild. 3 - 5 points: Moderate. 6 - 10 points: Severe.
SGRQ（St. George's Respiratory Questionnaire）Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  The SGRQ is used to evaluate the quality of life of patients with chronic respiratory diseases. It consists of three parts: symptoms, activities, and impact on daily life. The scoring range is 0 - 100 points. The higher the total score, the poorer the patient's quality of life.
mMRC（Modified Medical Research Council Dyspnea Scale）Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  The mMRC Score is used to assess the severity of dyspnoea and is divided into grades 0 - 4. The higher the score, the more severe the dyspnoea.
  Grade 0: Dyspnoea occurs only during strenuous exercise. Grade 1: Dyspnoea occurs when walking fast on flat ground or climbing a gentle slope.
  Grade 2: Dyspnoea causes the patient to stop and rest when walking on flat ground.
  Grade 3: Dyspnoea causes the patient to stop and rest after walking less than 100 metres or for a few minutes on flat ground.
  Grade 4: The patient is unable to leave home due to dyspnoea, or dyspnoea occurs when dressing or undressing.
ACT（Asthma Control Test） Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  The ACT Score is used to evaluate the quality of life of asthma patients in groups other than the chronic airway inflammation ICS research group. The scoring range is 5 - 25 points.
  Grade division:
  20 - 25 points: Asthma is well - controlled. 16 - 19 points: Asthma is partially - controlled. Less than 16 points: Asthma is uncontrolled.
AQLQ（Asthma Quality of Life Questionnaire）Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  The Asthma Quality of Life Questionnaire is used to evaluate the quality of life of asthma patients. The scoring range is 1 - 7 points. The higher the score, the better the quality of life.
FACED Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  FACED Score includes Forced Expiratory Volume in 1 second (FEV1)、Age、Chronic colonization by Pseudomonas aeruginosa (PA)、Extension (number of pulmonary lobes affected)、Dyspnea (mMRC score).It is used to assess the severity of bronchiectasis. The scoring range is from 0 to 10 points.
  Grade classification:
  0 - 2 points: Mild. 3 - 5 points: Moderate. 6 - 10 points: Severe.
BEST（Bronchiectasis Evaluation Score for Treatment)）Score | Baseline, Week 4 , Week 8 , and 3-month follow-up.
  The BEST Score is used to assess the symptoms of dyspnea and cough. The scoring range is from 0 to 10 points.
  Grade classification:
  0 - 2 points: Mild. 3 - 5 points: Moderate. 6 - 10 points: Severe.

IPD SHARING:
Plan to Share IPD: No